CLINICAL TRIAL: NCT01927094
Title: The Effect of a Probiotic and/or Prebiotic on the Duration of Diarrhea and Length of Hospital Stay in Children With Acute Diarrhea: Prospective, Double Blind, Randomized Controlled Trial
Brief Title: Effects of Probiotics and/or Prebiotics on the Duration of Diarrhea and Hospitalization in Children
Acronym: PROBAGE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Ener Cagri DINLEYICI, Associate Professor in Pediatrics, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROBAGE
Record Dates: First submitted 2013-08-13; First posted 2013-08-22 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Acute Diarrhea
Keywords: probiotics, diarrhea
MeSH Terms: conditions — Diarrhea | interventions — Probiotics; ORALIT

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic (Active Comparator): Saccharomyces boulardii 1 x 250 mg per day for 5 days, PO or Lactobacillus GG 1 x 10(9) CFU per day for 5 days or
  Lactobacillus reuteri 1 x 10(8) CFU per day for 5 days
  Interventions: Dietary Supplement: ORS
- Control (Active Comparator): ORS-ad libitum
  Interventions: Dietary Supplement: Probiotic

INTERVENTIONS:
Dietary Supplement: Probiotic — Comparison of probiotics vs. ORS
  Arms: Control
Dietary Supplement: ORS — ORS ad libitum
  Arms: Probiotic

SUMMARY:
* Acute diarrhea continues to be a major cause of childhood morbidity and mortality in developed and developing countries.
* Prevention and treatment of dehydration are the mainstays of therapy. Rehydration can be achieved with oral rehydratation solution (ORS).
* Even though ORS has reduced the mortality and morbidity very significantly, it has no effect on the duration of diarrhea, stool consistency and frequency and remains underused.
* ESPGHAN and ESPID published together an evidence based guideline and stated that in the management of acute gastroenteritis rehydration is the key treatment and that selected probiotics may reduce the duration and intensity of symptoms and can be used as an adjuvant to ORS.
* Current evidence also indicates that probiotic effects are strain-specific. Lactobacillus GG and Saccharomyces boulardii are the best studied strains. However, more research is needed to guide the use of particular probiotic regimens and strains and as there is still no evidence of efficacy for many preparations.

DETAILED DESCRIPTION:
Acute diarrhea continues to be a major cause of childhood morbidity and mortality in developed and developing countries. Prevention and treatment of dehydration are the mainstays of therapy. Rehydration can be achieved with oral rehydratation solution (ORS). Even though ORS has reduced the mortality and morbidity very significantly, it has no effect on the duration of diarrhea, stool consistency and frequency and remains underused. ESPGHAN and ESPID published together an evidence based guideline and stated that in the management of acute gastroenteritis rehydration is the key treatment and that selected probiotics may reduce the duration and intensity of symptoms and can be used as an adjuvant to ORS. A recent Cochrane review including 56 trials in children concluded that speciﬁc probiotics reduce the duration of diarrhea with about 24 hours and decrease the frequency of defecation on the second day. Current evidence also indicates that probiotic effects are strain-specific. Lactobacillus LGG and Saccharomyces boulardii are the best studied strains. However, more research is needed to guide the use of particular probiotic regimens and strains and as there is still no evidence of efficacy for many preparations. The aim of this study was to evaluate effects of different probiotics on the duration of acute infectious diarrhea.

ELIGIBILITY:
Inclusion Criteria:

* children of both sexes aged between 3 and 60 months, with acute watery diarrhea lasting more than 12 hours but less than 72 hours, requiring hospitalization. Children with clinical signs of mild to moderate dehydration (prolonged capillary refill time, abnormal skin turgor and 3-9% percentage loss of body weight).

Exclusion Criteria:

* clinical features of hypovolemic shock and/or necessitating admission at the intensive care unit were excluded. Other exclusion criteria were use of antibiotics or probiotics 1 month before admission, severe malnutrition and chronic underlying disease including immunocompromised conditions

Ages: 3 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1280 (Actual)
Dates: Start 2012-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Duration of diarrhea | Day 7
  Duration of diarrhea, since the beginning of the intervention, evaluated with Bristol scoring scale

SECONDARY OUTCOMES:
Percentage of children with diarrhea at the 3rd day of intervention | Day 3
  Percentage of children with diarrhea at the 3rd day of intervention
Duration of hospitalization | Day 5
  Lenght of stay of hoospitalization
Safety of probiotics | 5 days of intervention
  All clinical conditions (related with probiotics) should be noted.

CONTACTS AND LOCATIONS:
Overall Officials: Ener C Dinleyici, MD, Principal Investigator — Eskisehir Osmangazi University
Locations (3):
- Turkey (Türkiye) (3):
  - Dr. Sami Ulus Research and Training Hospital of Women's and Children's Health and Diseases, Ankara
  - Sisli Etfal Training and Research Hospital,, Istanbul
  - Umraniye Education & Research Hospital, Department of Pediatrics, Istanbul